CLINICAL TRIAL: NCT00256854
Title: A 4-Week, Randomized, Double-Blind, Cohort Study to Evaluate the Safety and Tolerability of Converting From Ropinirole Immediate Release (IR) to Ropinirole Controlled Release for RLS (CR-RLS) Formulation (Formerly Ropinirole Extended Release [XR]) in Patients With Restless Legs Syndrome (RLS)
Brief Title: Converting From Ropinirole Immediate Release (IR) To Ropinirole Controlled-Release for RLS (Restless Legs Syndrome)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: ROX104805
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2018-11

CONDITIONS: Restless Legs Syndrome; Restless Legs Syndrome (RLS)
Keywords: RLS; Ropinirole; Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — ropinirole

ARMS (6):
- Ropinirole cohort A1: 1 mg IR/2 mg CR-RLS/1 mg IR/1 mg IR (Experimental): Participants received Placebo in the evening and Ropinirole 1 mg IR at bedtime on Week 1. At the end of Week 1, participants were switched to receive Ropinirole 2 mg controlled release for Restless Legs Syndrome (CR-RLS) in the evening and placebo at bedtime till the end of Week 2. At the end of Week 2, participants were converted back to receive placebo in the evening and Ropinirole 1 mg IR at bedtime and continued to receive the same till the end of Week 4.
  Interventions: Drug: Ropinirole IR 1 mg; Drug: Ropinirole IR 1 mg Placebo; Drug: Ropinirole CR 2 mg; Drug: Ropinirole CR 2 mg Placebo
- Ropinirole cohort A2: 1 mg IR/1 mg IR/1 mg IR/2 mg CR-RLS (Experimental): Participants received Placebo in the evening and Ropinirole 1 mg IR at bedtime on Week 1 and continued to receive the same till the end of Week 3. At the end of Week 3, participants were switched to receive Ropinirole 2 mg CR-RLS in the evening and placebo at bedtime till the end of Week 4.
  Interventions: Drug: Ropinirole IR 1 mg; Drug: Ropinirole IR 1 mg Placebo; Drug: Ropinirole CR 2 mg; Drug: Ropinirole CR 2 mg Placebo
- Ropinirole cohort B1: 2 mg IR/3 mg CR-RLS/2 mg IR/2 mg IR (Experimental): Participants received Placebo in the evening and Ropinirole 2 mg IR at bedtime on Week 1. At the end of Week 1, participants were switched to receive Ropinirole 3 mg CR-RLS in the evening and placebo at bedtime till the end of Week 2. At the end of Week 2, participants were converted back to receive placebo in the evening and Ropinirole 2 mg IR at bedtime and continued to receive the same till the end of Week 4.
  Interventions: Drug: Ropinirole IR 2 mg; Drug: Ropinirole IR 2 mg Placebo; Drug: Ropinirole CR 3 mg; Drug: Ropinirole CR 3 mg Placebo
- Ropinirole cohort B2: 2 mg IR/2 mg IR/2 mg IR/3 mg CR-RLS (Experimental): Participants received Placebo in the evening and Ropinirole 2 mg IR at bedtime on Week 1 and continued to receive the same till the end of Week 3. At the end of Week 3, participants were switched to receive Ropinirole 3 mg CR-RLS in the evening and placebo at bedtime till the end of Week 4.
  Interventions: Drug: Ropinirole IR 2 mg; Drug: Ropinirole IR 2 mg Placebo; Drug: Ropinirole CR 3 mg; Drug: Ropinirole CR 3 mg Placebo
- Ropinirole cohort C1: 4 mg IR/6 mg CR-RLS/4 mg IR/4 mg IR (Experimental): Participants received Placebo in the evening and Ropinirole 4 mg IR at bedtime on Week 1. At the end of Week 1, participants were switched to receive Ropinirole 6 mg CR-RLS in the evening and placebo at bedtime till the end of Week 2. At the end of Week 2, participants were converted back to receive placebo in the evening and Ropinirole 4 mg IR at bedtime and continued to receive the same till the end of Week 4.
  Interventions: Drug: Ropinirole IR 2 mg; Drug: Ropinirole IR 2 mg Placebo; Drug: Ropinirole CR 3 mg; Drug: Ropinirole CR 3 mg Placebo
- Ropinirole cohort C2: 4 mg IR/4 mg IR/4 mg IR/6 mg CR-RLS (Experimental): Participants received Placebo in the evening and Ropinirole 4 mg IR at bedtime on Week 1 and continued to receive the same till the end of Week 3. At the end of Week 3, participants were switched to receive Ropinirole 6 mg CR-RLS in the evening and placebo at bedtime till the end of Week 4.
  Interventions: Drug: Ropinirole IR 2 mg; Drug: Ropinirole IR 2 mg Placebo; Drug: Ropinirole CR 3 mg; Drug: Ropinirole CR 3 mg Placebo

INTERVENTIONS:
Drug: Ropinirole IR 1 mg — Ropinirole IR (SKF-101468) will be supplied in the form of a 7mm round bi-convex white film coated tablet, de-bossed with 'GS' on both faces, containing ropinirole hydrochloride equivalent to 1.0mg of active drug substance.
  Other Names: ropinirole controlled-release for RLS
  Arms: Ropinirole cohort A1: 1 mg IR/2 mg CR-RLS/1 mg IR/1 mg IR; Ropinirole cohort A2: 1 mg IR/1 mg IR/1 mg IR/2 mg CR-RLS
Drug: Ropinirole IR 2 mg — Ropinirole IR (SKF-101468) will be supplied in the form of a 7mm round bi-convex white film coated tablet, de-bossed with 'GS' on both faces, containing ropinirole hydrochloride equivalent to 2.0mg of active drug substance.
  Arms: Ropinirole cohort B1: 2 mg IR/3 mg CR-RLS/2 mg IR/2 mg IR; Ropinirole cohort B2: 2 mg IR/2 mg IR/2 mg IR/3 mg CR-RLS; Ropinirole cohort C1: 4 mg IR/6 mg CR-RLS/4 mg IR/4 mg IR; Ropinirole cohort C2: 4 mg IR/4 mg IR/4 mg IR/6 mg CR-RLS
Drug: Ropinirole IR 1 mg Placebo — Ropinirole IR (SKF-101468) placebo will be supplied in the form of a 7mm round bi-convex white film coated tablet, de-bossed with 'GS' on both faces, containing matching placebo tablets of 1 mg.
  Arms: Ropinirole cohort A1: 1 mg IR/2 mg CR-RLS/1 mg IR/1 mg IR; Ropinirole cohort A2: 1 mg IR/1 mg IR/1 mg IR/2 mg CR-RLS
Drug: Ropinirole IR 2 mg Placebo — Ropinirole IR (SKF-101468) placebo will be supplied in the form of a 7mm round bi-convex white film coated tablet, de-bossed with 'GS' on both faces, containing matching placebo tablets of 2 mg.
  Arms: Ropinirole cohort B1: 2 mg IR/3 mg CR-RLS/2 mg IR/2 mg IR; Ropinirole cohort B2: 2 mg IR/2 mg IR/2 mg IR/3 mg CR-RLS; Ropinirole cohort C1: 4 mg IR/6 mg CR-RLS/4 mg IR/4 mg IR; Ropinirole cohort C2: 4 mg IR/4 mg IR/4 mg IR/6 mg CR-RLS
Drug: Ropinirole CR 2 mg — Ropinirole CR Tablets are presented as 7 mm round, bi-convex, white film coated tablets, de-bossed with 'GS' on both faces, containing ropinirole hydrochloride equivalent to 2mg of the active drug substance.
  Arms: Ropinirole cohort A1: 1 mg IR/2 mg CR-RLS/1 mg IR/1 mg IR; Ropinirole cohort A2: 1 mg IR/1 mg IR/1 mg IR/2 mg CR-RLS
Drug: Ropinirole CR 3 mg — Ropinirole CR Tablets are presented as 7 mm round, bi-convex, white film coated tablets, de-bossed with 'GS' on both faces, containing ropinirole hydrochloride equivalent to 3mg of the active drug substance.
  Arms: Ropinirole cohort B1: 2 mg IR/3 mg CR-RLS/2 mg IR/2 mg IR; Ropinirole cohort B2: 2 mg IR/2 mg IR/2 mg IR/3 mg CR-RLS; Ropinirole cohort C1: 4 mg IR/6 mg CR-RLS/4 mg IR/4 mg IR; Ropinirole cohort C2: 4 mg IR/4 mg IR/4 mg IR/6 mg CR-RLS
Drug: Ropinirole CR 2 mg Placebo — Ropinirole CR placebo Tablets are presented as 7 mm round, bi-convex, white film coated tablets, de-bossed with 'GS' on both faces, containing matching placebo tablets of 2 mg.
  Arms: Ropinirole cohort A1: 1 mg IR/2 mg CR-RLS/1 mg IR/1 mg IR; Ropinirole cohort A2: 1 mg IR/1 mg IR/1 mg IR/2 mg CR-RLS
Drug: Ropinirole CR 3 mg Placebo — Ropinirole CR placebo Tablets are presented as 7 mm round, bi-convex, white film coated tablets, de-bossed with 'GS' on both faces, containing matching placebo tablets of 3 mg.
  Arms: Ropinirole cohort B1: 2 mg IR/3 mg CR-RLS/2 mg IR/2 mg IR; Ropinirole cohort B2: 2 mg IR/2 mg IR/2 mg IR/3 mg CR-RLS; Ropinirole cohort C1: 4 mg IR/6 mg CR-RLS/4 mg IR/4 mg IR; Ropinirole cohort C2: 4 mg IR/4 mg IR/4 mg IR/6 mg CR-RLS

SUMMARY:
This is a multi-center, Phase III study to evaluate the safety and tolerability of proposed dose conversion recommendations for RLS subjects converting from ropinirole immediate release to ropinirole controlled-release for RLS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RLS using IRLS Study Group (IRLSSG) diagnostic criteria.
* Subjects currently being treated for RLS with a stable dose (for at least 2 weeks) of ropinirole IR given once daily.
* Subjects with RLS symptoms during both the evening and night or night time only.
* Subjects who have given written informed consent to participate.

Exclusion Criteria:

* Subjects who require treatment of daytime RLS symptoms.
* Signs of secondary RLS, serum ferritin level less than 10 mcg/L.
* Movement Disorders, Clinically significant or unstable medical conditions.
* Abnormal labs, electrocardiogram (ECG) or physical findings.
* Receiving prohibited medications.
* Sleeping habits incompatible with study design.
* Intolerance to ropinirole or other dopamine agonist.
* Pregnant or lactating.
* Women of child-bearing potential who are not practicing an acceptable method of birth control.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2005-11-14 (Actual); Primary Completion 2006-09-21 (Actual); Study Completion 2006-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- United States (30):
  - GSK Investigational Site, Laguna Hills, California
  - GSK Investigational Site, Oxnard, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Reseda, California
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Oak Brook, Illinois
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Bingham Farms, Michigan
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Cherry Hill, New Jersey
  - GSK Investigational Site, Toms River, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Plainview, New York
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Walla Walla, Washington
  - GSK Investigational Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: ROX104805 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: ROX104805 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: ROX104805 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: ROX104805 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: ROX104805 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: ROX104805 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: ROX104805 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 14 November 2005 till 21 September 2006 across 27 centers in the United States (US).
Pre-assignment Details: Participants with RLS were screened for 1 week; however, it could had been extended maximum up to 4 weeks. During screening period, participants received Ropinirole immediate release (IR) 1 milligrams (mg), 2 mg, or 4 mg across Cohorts A, B, and C. A total of 135 participants were randomized in the study.
Period: Overall Study
Arm/Group | Ropinirole Cohort A1: 1 mg IR/2 mg CR-RLS/1 mg IR/1 mg IR | Ropinirole Cohort A2: 1 mg IR/1 mg IR/1 mg IR/2 mg CR-RLS | Ropinirole Cohort B1: 2 mg IR/3 mg CR-RLS/2 mg IR/2 mg IR | Ropinirole Cohort B2: 2 mg IR/2 mg IR/2 mg IR/3 mg CR-RLS | Ropinirole Cohort C1: 4 mg IR/6 mg CR-RLS/4 mg IR/4 mg IR | Ropinirole Cohort C2: 4 mg IR/4 mg IR/4 mg IR/6 mg CR-RLS
Started | 26 | 26 | 26 | 27 | 16 | 14
Completed | 23 | 22 | 23 | 24 | 15 | 13
Not Completed | 3 | 4 | 3 | 3 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 3 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 2 | 0 | 1
Not completed — Not compliant with the study drug | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who entered into the study and who received at least one dose of the double-blind medication.
Groups:
- Ropinirole Cohort A1: 1 mg IR/2 mg CR-RLS/1 mg IR/1 mg IR: Participants received Placebo in the evening and Ropinirole 1 mg IR at bedtime on Week 1. At the end of Week 1, participants were switched to receive Ropinirole 2 mg CR-RLS in the evening and placebo at bedtime till the end of Week 2. At the end of Week 2, participants were converted back to receive placebo in the evening and Ropinirole 1 mg IR at bedtime and continued to receive the same till the end of Week 4.
- Total: Total of all reporting groups
Arm/Group | Ropinirole Cohort A1: 1 mg IR/2 mg CR-RLS/1 mg IR/1 mg IR | Ropinirole Cohort A2: 1 mg IR/1 mg IR/1 mg IR/2 mg CR-RLS | Ropinirole Cohort B1: 2 mg IR/3 mg CR-RLS/2 mg IR/2 mg IR | Ropinirole Cohort B2: 2 mg IR/2 mg IR/2 mg IR/3 mg CR-RLS | Ropinirole Cohort C1: 4 mg IR/6 mg CR-RLS/4 mg IR/4 mg IR | Ropinirole Cohort C2: 4 mg IR/4 mg IR/4 mg IR/6 mg CR-RLS | Total
Number analyzed (Participants) | 26 | 26 | 26 | 27 | 16 | 14 | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.8 (12.91) | 57.4 (8.69) | 59.2 (10.21) | 53.7 (13.94) | 58.3 (11.96) | 57.1 (9.67) | 57.0 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 14 | 18 | 7 | 7 | 84
  Male | 6 | 8 | 12 | 9 | 9 | 7 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 1 | 0 | 3
  White | 25 | 24 | 25 | 27 | 15 | 14 | 130
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) Post-conversion From Ropinirole IR to Ropinirole CR Over Period
Description: AE is an unfavorable change in the health of a participant, including abnormal laboratory findings, that happens during a clinical study or within a certain time period after the study has ended. This change may or may not be caused by the intervention being studied. In each of the 6 cohorts, there were 2 conversions, one of which was IR to CR-RLS and the other one IR to IR. Two populations were defined: the first conversion population and the second conversion population. The first conversion population consisted of all participants receiving at least one dose of randomized drug during the pre-conversion 1 period and during the post-conversion 1 period. The second conversion population consisted of all participants receiving at least one dose of randomized drug during the pre-conversion 2 period and during the post-conversion 2 period.
Time Frame: Up to 5 weeks
Population: Conversion population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Ropinirole Cohort A1: 1 mg IR/2 mg CR-RLS/1 mg IR/1 mg IR | Ropinirole Cohort A2: 1 mg IR/1 mg IR/1 mg IR/2 mg CR-RLS | Ropinirole Cohort B1: 2 mg IR/3 mg CR-RLS/2 mg IR/2 mg IR | Ropinirole Cohort B2: 2 mg IR/2 mg IR/2 mg IR/3 mg CR-RLS | Ropinirole Cohort C1: 4 mg IR/6 mg CR-RLS/4 mg IR/4 mg IR | Ropinirole Cohort C2: 4 mg IR/4 mg IR/4 mg IR/6 mg CR-RLS
Number analyzed (Participants) | 24 | 24 | 26 | 26 | 15 | 13
Participants
  Post-conversion 1 | 9 | 14 | 10 | 11 | 7 | 5
  Post-conversion 2: number analyzed (Participants) | 23 | 22 | 23 | 24 | 15 | 13
  Post-conversion 2 | 6 | 8 | 7 | 6 | 5 | 6

2. Secondary Outcome: Number of Participants Discontinuing the Drug Due to AEs Post Conversion From Ropinirole IR to Ropinirole CR-RLS
Description: AE is an unfavorable change in the health of a participant, including abnormal laboratory findings, that happens during a clinical study or within a certain time period after the study has ended. This change may or may not be caused by the intervention being studied. Onset of an AE was pre-Conversion 1 and discontinuation for the same AE occurred post-Conversion 1. Serious adverse event (SAE) is an adverse event that results in death, is life-threatening, requires inpatient hospitalization or extends a current hospital stay, results in an ongoing or significant incapacity or interferes substantially with normal life functions, or causes a congenital anomaly or birth defect. Medical events that do not result in death, are not life-threatening, or do not require hospitalization may be considered serious adverse events if they put the participant in danger or require medical or surgical intervention to prevent one of the results listed above.
Time Frame: Up to 5 weeks
Population: Conversion population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Ropinirole Cohort A1: 1 mg IR/2 mg CR-RLS/1 mg IR/1 mg IR | Ropinirole Cohort A2: 1 mg IR/1 mg IR/1 mg IR/2 mg CR-RLS | Ropinirole Cohort B1: 2 mg IR/3 mg CR-RLS/2 mg IR/2 mg IR | Ropinirole Cohort B2: 2 mg IR/2 mg IR/2 mg IR/3 mg CR-RLS | Ropinirole Cohort C1: 4 mg IR/6 mg CR-RLS/4 mg IR/4 mg IR | Ropinirole Cohort C2: 4 mg IR/4 mg IR/4 mg IR/6 mg CR-RLS
Number analyzed (Participants) | 24 | 24 | 26 | 26 | 15 | 13
Participants
  Post-conversion 1 | 0 | 0 | 1 | 1 | 0 | 0
  Post-conversion 2: number analyzed (Participants) | 23 | 22 | 23 | 24 | 15 | 13
  Post-conversion 2 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With SAEs and Severity of AEs
Description: SAE is an adverse event that results in death, is life-threatening, requires inpatient hospitalization or extends a current hospital stay, results in an ongoing or significant incapacity or interferes substantially with normal life functions, or causes a congenital anomaly or birth defect. Medical events that do not result in death, are not life-threatening, or do not require hospitalization may be considered serious adverse events if they put the participant in danger or require medical or surgical intervention to prevent one of the results listed above. Severity was measured in terms of grades mild, moderate, and severe. SAEs data only for post-conversion has been reported.
Time Frame: Up to 5 weeks
Population: Conversion population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Ropinirole Cohort A1: 1 mg IR/2 mg CR-RLS/1 mg IR/1 mg IR | Ropinirole Cohort A2: 1 mg IR/1 mg IR/1 mg IR/2 mg CR-RLS | Ropinirole Cohort B1: 2 mg IR/3 mg CR-RLS/2 mg IR/2 mg IR | Ropinirole Cohort B2: 2 mg IR/2 mg IR/2 mg IR/3 mg CR-RLS | Ropinirole Cohort C1: 4 mg IR/6 mg CR-RLS/4 mg IR/4 mg IR | Ropinirole Cohort C2: 4 mg IR/4 mg IR/4 mg IR/6 mg CR-RLS
Number analyzed (Participants) | 24 | 24 | 26 | 26 | 15 | 13
Participants
  Any SAE, post conversion 1 | 0 | 0 | 0 | 0 | 0 | 0
  Any SAE, post conversion 2: number analyzed (Participants) | 23 | 22 | 23 | 24 | 15 | 13
  Any SAE, post conversion 2 | 0 | 0 | 0 | 0 | 0 | 0
  Mild AE, post conversion 1 | 5 | 9 | 5 | 6 | 3 | 2
  Moderate AE, post conversion 1 | 4 | 7 | 4 | 6 | 4 | 4
  Severe AE, post conversion 1 | 2 | 5 | 6 | 2 | 2 | 1
  Mild AE, post conversion 2: number analyzed (Participants) | 23 | 22 | 23 | 24 | 15 | 13
  Mild AE, post conversion 2 | 3 | 2 | 1 | 1 | 2 | 1
  Moderate AE, post conversion 2: number analyzed (Participants) | 23 | 22 | 23 | 24 | 15 | 13
  Moderate AE, post conversion 2 | 2 | 4 | 3 | 5 | 4 | 1
  Severe AE, post conversion 2: number analyzed (Participants) | 23 | 22 | 23 | 24 | 15 | 13
  Severe AE, post conversion 2 | 2 | 2 | 3 | 0 | 0 | 4

4. Secondary Outcome: Number of Participants With Positive Scores (Improved) on Clinical Global Impression Improvement Scale (CGI-I) Pre-conversion and One Week Post-conversion
Description: Global Improvement Scale (CGI-I) allows the Investigator to rate the participants' global improvement or worsening compared with the condition at Baseline (Day 0), whether or not the change is thought to be due to treatment with study drug. The scale is rated from 1 to 7 (1="Very much improved" to 7="Very much worse"). Typically, a participant with a score of 1 were considered as "Very much improved" and 2 as "Much improved" responder. Positive response was given in terms of worsen to stable or stable to improved.
Time Frame: Up to 4 weeks
Population: First and Second Conversion Populations. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Ropinirole Cohort A1: 1 mg IR/2 mg CR-RLS/1 mg IR/1 mg IR | Ropinirole Cohort A2: 1 mg IR/1 mg IR/1 mg IR/2 mg CR-RLS | Ropinirole Cohort B1: 2 mg IR/3 mg CR-RLS/2 mg IR/2 mg IR | Ropinirole Cohort B2: 2 mg IR/2 mg IR/2 mg IR/3 mg CR-RLS | Ropinirole Cohort C1: 4 mg IR/6 mg CR-RLS/4 mg IR/4 mg IR | Ropinirole Cohort C2: 4 mg IR/4 mg IR/4 mg IR/6 mg CR-RLS
Number analyzed (Participants) | 24 | 24 | 26 | 26 | 15 | 13
Participants
  Post Coversion 1: number analyzed (Participants) | 24 | 24 | 24 | 23 | 15 | 13
  Post Coversion 1 | 14 | 12 | 10 | 9 | 6 | 6
  Post Conversion 2: number analyzed (Participants) | 23 | 21 | 23 | 23 | 14 | 13
  Post Conversion 2 | 11 | 14 | 13 | 14 | 5 | 7

5. Secondary Outcome: Change From Pre-conversion in International RLS (IRLS) Rating Scale Total Score to One Week Post-conversion
Description: The IRLS Rating Scale was developed to measure disease severity for clinical assessment, research, and therapeutic studies an also to show relationship between responses and overall RLS severity. The IRLS Rating Scale is a disease-specific 10-item scale that is based on the IRLSSG consensus of clinical features and associated sleep problems. The investigator asked the participant to rate his/her symptoms for each of the ten questions contained in the IRLS Rating Scale from 0 to 4, with 0 representing the absence of a problem and 4 a very severe problem. The best and worst possible scores are 0 and 40, respectively; higher scores represent a greater severity of symptoms. Changes from pre- to one-week post-conversion in the IRLS rating scale total score was obtained by subtracting the "Week 1" total score from the "Week 2" total score for the first conversion and the "Week 3" total score from the "Week 4" total score for the second conversion.
Time Frame: Up to 5 weeks
Population: Conversion populations. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ropinirole Cohort A1: 1 mg IR/2 mg CR-RLS/1 mg IR/1 mg IR | Ropinirole Cohort A2: 1 mg IR/1 mg IR/1 mg IR/2 mg CR-RLS | Ropinirole Cohort B1: 2 mg IR/3 mg CR-RLS/2 mg IR/2 mg IR | Ropinirole Cohort B2: 2 mg IR/2 mg IR/2 mg IR/3 mg CR-RLS | Ropinirole Cohort C1: 4 mg IR/6 mg CR-RLS/4 mg IR/4 mg IR | Ropinirole Cohort C2: 4 mg IR/4 mg IR/4 mg IR/6 mg CR-RLS
Number analyzed (Participants) | 24 | 24 | 26 | 26 | 15 | 13
Scores on a scale
  Post-Conversion 1: number analyzed (Participants) | 24 | 24 | 24 | 23 | 15 | 13
  Post-Conversion 1 | -5.1 (8.84) | -0.1 (7.34) | -1.5 (6.73) | -1.3 (7.15) | -5.8 (6.14) | 1.2 (10.33)
  Post-Conversion 2: number analyzed (Participants) | 23 | 21 | 23 | 23 | 14 | 13
  Post-Conversion 2 | -2.9 (7.07) | -4.8 (7.73) | -1.6 (6.29) | -5.2 (9.62) | 0.6 (7.28) | -2.2 (11.58)

6. Secondary Outcome: Number of Participants With pre-and One Week Post-conversion Values of Vital Signs of Potential Clinical Concern (PCC)
Description: The number of participants with pre- and post- conversion orthostatic systolic blood pressure (SBP), diastolic blood pressure (DBP) and pulse rate values of PCC were summarized. Both conversions (drug and dummy) were considered. High and low values of only orthostatic SBP and DBP of PCC are presented.
Time Frame: Up to 5 weeks
Population: Conversion populations. Only those participants at the indicated conversion were analyzed. The population from Cohort A1 and A2 are pooled to a single arm Cohort A. Similarly populations B1, B2 and C1, C2 are pooled to Cohort B and Cohort C, respectively.
Measure: Count of Participants; unit: Participants
Groups:
- Ropinirole Cohort A: It consisted of two dosing groups: A1 and A2. In cohort A1, participants received Placebo in the evening and Ropinirole 1mg IR at bedtime on Week 1. At the end of Week 1, participants were switched to receive Ropinirole 2 mg CR-RLS in the evening and placebo at bedtime till the end of Week 2. At the end of Week 2, participants were converted back to receive placebo in the evening and Ropinirole 1 mg IR at bedtime and continued to receive the same till the end of Week 4. In cohort A2, participants received Placebo in the evening and Ropinirole 1 mg IR at bedtime on Week 1 and continued to receive the same till the end of Week 3. At the end of Week 3, participants were switched to receive Ropinirole 2 mg CR-RLS in the evening and placebo at bedtime till the end of Week 4.
- Ropinirole Cohort B: It consisted of two dosing groups: B1 and B2. In cohort B1, participants received Placebo in the evening and Ropinirole 2 mg IR at bedtime on Week 1. At the end of Week 1, participants were switched to receive Ropinirole 3 mg CR-RLS in the evening and placebo at bedtime till the end of Week 2. At the end of Week 2, participants were converted back to receive placebo in the evening and Ropinirole 2 mg IR at bedtime and continued to receive the same till the end of Week 4. In cohort B2, participants received Placebo in the evening and Ropinirole 2 mg IR at bedtime on Week 1 and continued to receive the same till the end of Week 3. At the end of Week 3, participants were switched to receive Ropinirole 3 mg CR-RLS in the evening and placebo at bedtime till the end of Week 4.
- Ropinirole Cohort C: It consisted of two dosing groups: C1 and C2. In cohort C1, participants received Placebo in the evening and Ropinirole 4 mg IR at bedtime on Week 1. At the end of Week 1, participants were switched to receive Ropinirole 6 mg CR-RLS in the evening and placebo at bedtime till the end of Week 2. At the end of Week 2, participants were converted back to receive placebo in the evening and Ropinirole 4 mg IR at bedtime and continued to receive the same till the end of Week 4. In cohort C2, participants received Placebo in the evening and Ropinirole 4 mg IR at bedtime on Week 1 and continued to receive the same till the end of Week 3. At the end of Week 3, participants were switched to receive Ropinirole 6 mg CR-RLS in the evening and placebo at bedtime till the end of Week 4.
Arm/Group | Ropinirole Cohort A | Ropinirole Cohort B | Ropinirole Cohort C
Number analyzed (Participants) | 52 | 53 | 30
Participants
  1 mg IR to 2 mg CR, SBP, PCC low, pre-conversion: number analyzed (Participants) | 46 | 0 | 0
  1 mg IR to 2 mg CR, SBP, PCC low, pre-conversion | 1 |  |
  1 mg IR to 1 mg IR, SBP, PCC high, post-conversion: number analyzed (Participants) | 47 | 0 | 0
  1 mg IR to 1 mg IR, SBP, PCC high, post-conversion | 1 |  |
  2 mg IR to 3 mg CR, SBP, PCC high, pre-conversion: number analyzed (Participants) | 0 | 46 | 0
  2 mg IR to 3 mg CR, SBP, PCC high, pre-conversion |  | 1 |
  2 mg IR to 2 mg IR,SBP, PCC high, post-conversion: number analyzed (Participants) | 0 | 47 | 0
  2 mg IR to 2 mg IR,SBP, PCC high, post-conversion |  | 1 |
  4 mg IR to 4 mg IR, SBP, PCC high, pre-conversion: number analyzed (Participants) | 0 | 0 | 28
  4 mg IR to 4 mg IR, SBP, PCC high, pre-conversion |  |  | 1
  1 mg IR to 2 mg CR, DBP, PCC high, pre-conversion: number analyzed (Participants) | 46 | 0 | 0
  1 mg IR to 2 mg CR, DBP, PCC high, pre-conversion | 2 |  |
  1 mg IR to 2 mg CR, DBP, PCC high, post-conversion: number analyzed (Participants) | 45 | 0 | 0
  1 mg IR to 2 mg CR, DBP, PCC high, post-conversion | 3 |  |
  1 mg IR to 1 mg IR, DBP, PCC high, pre-conversion: number analyzed (Participants) | 47 | 0 | 0
  1 mg IR to 1 mg IR, DBP, PCC high, pre-conversion | 4 |  |
  1 mg IR to 1 mg IR, DBP, PCC high, post-conversion: number analyzed (Participants) | 47 | 0 | 0
  1 mg IR to 1 mg IR, DBP, PCC high, post-conversion | 2 |  |
  2 mg IR to 3 mg CR, DBP, PCC high, pre-conversion: number analyzed (Participants) | 0 | 46 | 0
  2 mg IR to 3 mg CR, DBP, PCC high, pre-conversion |  | 1 |
  2 mg IR to 3 mg CR, DBP, PCC high, post-conversion: number analyzed (Participants) | 0 | 45 | 0
  2 mg IR to 3 mg CR, DBP, PCC high, post-conversion |  | 6 |
  2 mg IR to 2 mg IR, DBP, PCC high, pre-conversion: number analyzed (Participants) | 0 | 47 | 0
  2 mg IR to 2 mg IR, DBP, PCC high, pre-conversion |  | 2 |
  2 mg IR to 2 mg IR, DBP, PCC high, post-conversion: number analyzed (Participants) | 0 | 47 | 0
  2 mg IR to 2 mg IR, DBP, PCC high, post-conversion |  | 2 |
  4 mg IR to 6 mg CR, DBP, PCC high, post-conversion: number analyzed (Participants) | 0 | 0 | 28
  4 mg IR to 6 mg CR, DBP, PCC high, post-conversion |  |  | 4
  4 mg IR to 4 mg IR, DBP, PCC high, pre-conversion: number analyzed (Participants) | 0 | 0 | 28
  4 mg IR to 4 mg IR, DBP, PCC high, pre-conversion |  |  | 1
  4 mg IR to 4 mg IR, DBP, PCC high, post-conversion: number analyzed (Participants) | 0 | 0 | 27
  4 mg IR to 4 mg IR, DBP, PCC high, post-conversion |  |  | 2
  1 mg IR to 1 mg IR, pulse, PCC low,post-conversion: number analyzed (Participants) | 47 | 0 | 0
  1 mg IR to 1 mg IR, pulse, PCC low,post-conversion | 1 |  |
  2 mg IR to 3 mg CR, pulse, PCC high,pre-conversion: number analyzed (Participants) | 0 | 46 | 0
  2 mg IR to 3 mg CR, pulse, PCC high,pre-conversion |  | 1 |
  2 mg IR to 2 mg IR, pulse,PCC high,post-conversion: number analyzed (Participants) | 0 | 47 | 0
  2 mg IR to 2 mg IR, pulse,PCC high,post-conversion |  | 2 |

7. Secondary Outcome: Change From Pre-conversion in Systolic and Diastolic Orthostatic SBP and DBP to One Week Post-conversion
Description: Both conversions 1 and 2 (drug and dummy) were considered for analysis. High and low values of only orthostatic SBP and DBP of PCC are presented. Change from pre-conversion in BP is the value of BP at post-conversion minus the value at pre-conversion. For orthostatic changes (standing minus semi-supine vital signs values), pre-conversion measurements were compared with the post-conversion measurements. Positive values are indicative of less orthostatic decrease in blood pressure. The first conversion relates to the Week 1 visit, with pre- to post-conversion changes computed as "Week 2" values minus the Week 1" values, and the second conversion relates to the Week 3 visit with pre- to post-conversion changes computed as the "Week 4" values minus the Week 3" values.
Time Frame: Up to 5 weeks
Population: Conversion Populations. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mm of Hg)
Arm/Group | Ropinirole Cohort A1: 1 mg IR/2 mg CR-RLS/1 mg IR/1 mg IR | Ropinirole Cohort A2: 1 mg IR/1 mg IR/1 mg IR/2 mg CR-RLS | Ropinirole Cohort B1: 2 mg IR/3 mg CR-RLS/2 mg IR/2 mg IR | Ropinirole Cohort B2: 2 mg IR/2 mg IR/2 mg IR/3 mg CR-RLS | Ropinirole Cohort C1: 4 mg IR/6 mg CR-RLS/4 mg IR/4 mg IR | Ropinirole Cohort C2: 4 mg IR/4 mg IR/4 mg IR/6 mg CR-RLS
Number analyzed (Participants) | 24 | 24 | 26 | 26 | 15 | 13
Millimeters of mercury (mm of Hg)
  Semi-supine SBP, conversion 1: number analyzed (Participants) | 24 | 24 | 24 | 23 | 15 | 13
  Semi-supine SBP, conversion 1 | -0.8 (12.08) | -3.9 (13.78) | 4.0 (10.81) | -7.7 (10.20) | -1.2 (7.85) | -5.3 (17.84)
  Standing SBP, conversion 1: number analyzed (Participants) | 24 | 24 | 24 | 22 | 15 | 13
  Standing SBP, conversion 1 | 2.3 (12.57) | -2.9 (13.18) | -0.2 (14.19) | -4.1 (10.75) | 0.7 (6.64) | -3.9 (11.43)
  Semi-supine SBP, conversion 2: number analyzed (Participants) | 23 | 21 | 23 | 23 | 14 | 13
  Semi-supine SBP, conversion 2 | 1.6 (14.51) | 0.6 (10.33) | 0.3 (8.91) | 2.1 (10.73) | -2.6 (8.81) | -6.2 (19.61)
  Standing SBP, conversion 2: number analyzed (Participants) | 23 | 21 | 23 | 23 | 14 | 13
  Standing SBP, conversion 2 | -0.3 (13.24) | 3.1 (14.59) | 3.6 (9.23) | 1.0 (12.90) | 0.4 (12.42) | -4.9 (16.82)
  Orhostatic SBP, post-conversion 1: number analyzed (Participants) | 24 | 24 | 24 | 22 | 15 | 13
  Orhostatic SBP, post-conversion 1 | 3.2 (10.69) | 1.0 (10.29) | -4.2 (12.12) | 3.4 (9.95) | 1.9 (7.76) | 1.4 (9.69)
  Orthostatic SBP, post-conversion 2: number analyzed (Participants) | 23 | 21 | 23 | 23 | 14 | 13
  Orthostatic SBP, post-conversion 2 | -1.9 (10.18) | 2.5 (13.32) | 3.3 (8.42) | -1.0 (9.73) | 3.0 (13.46) | 1.3 (12.39)
  Semi-supine DBP, conversion 1: number analyzed (Participants) | 24 | 24 | 24 | 23 | 15 | 13
  Semi-supine DBP, conversion 1 | 1.3 (10.96) | -2.5 (8.10) | 2.2 (10.43) | -3.5 (6.52) | -1.3 (7.61) | -1.2 (6.91)
  Standing DBP, conversion 1: number analyzed (Participants) | 24 | 24 | 24 | 22 | 15 | 13
  Standing DBP, conversion 1 | 3.3 (7.56) | -3.4 (10.25) | 4.1 (11.45) | -3.2 (7.11) | 0.6 (6.07) | -0.8 (10.08)
  Semi-supine DBP, conversion 2: number analyzed (Participants) | 23 | 24 | 23 | 23 | 14 | 13
  Semi-supine DBP, conversion 2 | -0.5 (8.67) | 2.8 (8.80) | 1.3 (5.53) | -0.7 (8.17) | 0.0 (5.45) | -0.7 (13.24)
  Standing DBP, conversion 2: number analyzed (Participants) | 23 | 24 | 23 | 23 | 14 | 13
  Standing DBP, conversion 2 | -2.7 (8.64) | 2.8 (7.92) | 0.3 (7.42) | 0.7 (8.91) | -0.3 (6.76) | 1.8 (12.14)
  Orthostatic DBP, post-conversion 1: number analyzed (Participants) | 24 | 24 | 24 | 22 | 15 | 13
  Orthostatic DBP, post-conversion 1 | 2.0 (7.22) | -0.9 (7.11) | 1.9 (9.70) | 0.5 (6.37) | 1.9 (6.53) | 0.4 (8.17)
  Orthostatic DBP, post-conversion 2: number analyzed (Participants) | 23 | 21 | 23 | 23 | 14 | 13
  Orthostatic DBP, post-conversion 2 | -2.2 (5.69) | 0.0 (6.30) | -1.1 (6.49) | 1.4 (7.82) | -0.3 (3.31) | 2.5 (8.37)

8. Secondary Outcome: Change From Pre-conversion in Pulse Rate to One Week Post-conversion
Description: Both conversions 1 and 2 (drug and dummy) were considered for analysis. High and low values of only orthostatic pulse of PCC are presented. Change from pre-conversion in pulse rate is the value of pulse rate at post-conversion minus the value at pre-conversion. For orthostatic changes (standing minus semi-supine vital signs values), pre-conversion measurements were compared with the post-conversion measurements. Positive values are indicative of less orthostatic decrease in pulse. The first conversion relates to the Week 1 visit, with pre- to post-conversion changes computed as "Week 2" values minus the "Week 1" values, and the second conversion relates to the Week 3 visit with pre- to post-conversion changes computed as the "Week 4" values minus the "Week 3" values.
Time Frame: Up to 5 weeks
Population: Conversion Populations. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Ropinirole Cohort A1: 1 mg IR/2 mg CR-RLS/1 mg IR/1 mg IR | Ropinirole Cohort A2: 1 mg IR/1 mg IR/1 mg IR/2 mg CR-RLS | Ropinirole Cohort B1: 2 mg IR/3 mg CR-RLS/2 mg IR/2 mg IR | Ropinirole Cohort B2: 2 mg IR/2 mg IR/2 mg IR/3 mg CR-RLS | Ropinirole Cohort C1: 4 mg IR/6 mg CR-RLS/4 mg IR/4 mg IR | Ropinirole Cohort C2: 4 mg IR/4 mg IR/4 mg IR/6 mg CR-RLS
Number analyzed (Participants) | 26 | 26 | 26 | 27 | 16 | 14
Beats per minute (bpm)
  Semi-supine pulse, Conversion 1: number analyzed (Participants) | 24 | 24 | 24 | 23 | 15 | 13
  Semi-supine pulse, Conversion 1 | -0.1 (7.01) | -0.4 (5.38) | 1.0 (9.42) | -0.9 (6.81) | -1.5 (6.99) | 1.2 (8.09)
  Standing pulse, Conversion 1: number analyzed (Participants) | 24 | 24 | 24 | 22 | 15 | 13
  Standing pulse, Conversion 1 | 2.4 (8.39) | 0.3 (9.48) | 0.0 (10.71) | 0.7 (8.82) | -0.8 (7.84) | -0.8 (8.69)
  Semi-supine pulse, Conversion 2: number analyzed (Participants) | 23 | 21 | 23 | 23 | 14 | 13
  Semi-supine pulse, Conversion 2 | -0.7 (8.11) | 0.3 (6.81) | 0.2 (9.05) | 0.3 (8.49) | 0.6 (5.18) | -0.8 (8.97)
  Standing pulse, Conversion 2: number analyzed (Participants) | 23 | 21 | 23 | 23 | 14 | 13
  Standing pulse, Conversion 2 | -0.4 (9.36) | 0.3 (8.95) | 1.4 (12.77) | 0.9 (9.01) | 0.9 (5.99) | 1.5 (8.53)
  Post-Conversion 1: number analyzed (Participants) | 24 | 24 | 24 | 22 | 15 | 13
  Post-Conversion 1 | 2.5 (8.80) | 0.7 (8.38) | -1.0 (6.72) | 1.6 (8.29) | 0.7 (4.59) | -2.0 (7.56)
  Post-Conversion 2: number analyzed (Participants) | 23 | 21 | 23 | 23 | 14 | 13
  Post-Conversion 2 | 0.3 (9.27) | 0.0 (6.78) | 1.2 (9.87) | 0.6 (6.24) | 0.3 (6.07) | 2.2 (5.37)

9. Secondary Outcome: Change From Pre-conversion to Post-conversion in Ambulatory Blood Pressure
Description: Blood pressure (both systolic and diastolic) measurements were made just prior to the first dose of study medication ('evening' dose, ropinirole CR-RLS or matching placebo) and then every hour afterwards up to bedtime (when the device was removed). The changes for the first conversion were calculated as the "post evening dose" values minus the "pre evening dose" values at the Week 1 visit and the changes for the second conversion were the "post evening dose" values minus the "pre evening dose" values at the Week 3 visit.
Time Frame: Up to 5 weeks
Population: Conversion population. Only those participants available at the time of conversion were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Ropinirole Cohort A1: 1 mg IR/2 mg CR-RLS/1 mg IR/1 mg IR: Participants received Placebo in the evening and Ropinirole 1 milligram (mg) immediate release (IR) at bedtime on Week 1. At the end of Week 1, participants were switched to receive Ropinirole 2 mg controlled release for Restless Legs Syndrome (CR-RLS) in the evening and placebo at bedtime till the end of Week 2. At the end of Week 2, participants were converted back to receive placebo in the evening and Ropinirole 1 mg IR at bedtime and continued to receive the same till the end of Week 4.
Arm/Group | Ropinirole Cohort A1: 1 mg IR/2 mg CR-RLS/1 mg IR/1 mg IR | Ropinirole Cohort A2: 1 mg IR/1 mg IR/1 mg IR/2 mg CR-RLS | Ropinirole Cohort B1: 2 mg IR/3 mg CR-RLS/2 mg IR/2 mg IR | Ropinirole Cohort B2: 2 mg IR/2 mg IR/2 mg IR/3 mg CR-RLS | Ropinirole Cohort C1: 4 mg IR/6 mg CR-RLS/4 mg IR/4 mg IR | Ropinirole Cohort C2: 4 mg IR/4 mg IR/4 mg IR/6 mg CR-RLS
Number analyzed (Participants) | 24 | 24 | 26 | 26 | 15 | 13
mmHg
  SBP, conversion 1, <30 minutes: number analyzed (Participants) | 1 | 0 | 1 | 1 | 0 | 0
  SBP, conversion 1, <30 minutes | -20.0 (NA) — only one participant was analyzed, hence SD was not calculated. |  | -20.0 (NA) — only one participant was analyzed, hence SD was not calculated. | -6.0 (NA) — only one participant was analyzed, hence SD was not calculated. |  |
  SBP, conversion 1, 1 hour: number analyzed (Participants) | 12 | 14 | 14 | 12 | 8 | 2
  SBP, conversion 1, 1 hour | -8.0 (10.64) | -6.4 (14.14) | -10.6 (9.86) | -1.0 (10.96) | -6.3 (8.35) | -5.0 (2.83)
  SBP, conversion 1, 2 hours: number analyzed (Participants) | 11 | 15 | 13 | 11 | 8 | 2
  SBP, conversion 1, 2 hours | -12.9 (14.10) | 0.1 (16.83) | -9.1 (6.84) | -4.3 (10.35) | -8.0 (7.19) | 7.5 (4.95)
  SBP, conversion 1, 3 hours: number analyzed (Participants) | 12 | 12 | 11 | 10 | 5 | 2
  SBP, conversion 1, 3 hours | -10.8 (13.57) | 1.3 (12.46) | -15.9 (13.71) | -3.0 (9.49) | -7.4 (8.82) | -4.5 (0.71)
  SBP, conversion 1, 4 hours: number analyzed (Participants) | 7 | 11 | 10 | 8 | 4 | 2
  SBP, conversion 1, 4 hours | -11.0 (7.26) | -9.9 (17.40) | -12.8 (15.82) | -10.3 (7.74) | -12.8 (12.89) | 3.5 (2.12)
  SBP, conversion 1, 5 hours: number analyzed (Participants) | 5 | 7 | 4 | 4 | 2 | 1
  SBP, conversion 1, 5 hours | -8.6 (7.70) | -10.6 (20.86) | -15.5 (13.77) | -8.3 (5.91) | -15.5 (6.36) | 14.0 (NA) — only one participant was analyzed, hence SD was not calculated.
  SBP, conversion 1, 6 hours: number analyzed (Participants) | 3 | 1 | 3 | 2 | 0 | 1
  SBP, conversion 1, 6 hours | -14.3 (4.51) | -11.0 (NA) — only one participant was analyzed, hence SD was not calculated. | -9.0 (21.38) | -11.0 (25.46) |  | 0.0 (NA) — only one participant was analyzed, hence SD was not calculated.
  SBP, conversion 2, <30 minutes: number analyzed (Participants) | 0 | 1 | 0 | 0 | 2 | 1
  SBP, conversion 2, <30 minutes |  | -15.0 (NA) — only one participant was analyzed, hence SD was not calculated. |  |  | -5.5 (4.95) | 12.0 (NA) — only one participant was analyzed, hence SD was not calculated.
  SBP, conversion 2, 1 hour: number analyzed (Participants) | 5 | 12 | 11 | 7 | 9 | 5
  SBP, conversion 2, 1 hour | -5.4 (11.35) | -1.5 (13.81) | -1.6 (9.80) | -1.3 (13.47) | 0.6 (10.71) | -2.8 (3.77)
  SBP, conversion 2, 2 hours: number analyzed (Participants) | 5 | 11 | 12 | 7 | 8 | 4
  SBP, conversion 2, 2 hours | 2.6 (19.23) | -10.6 (17.44) | 2.0 (6.62) | -0.6 (16.33) | -0.3 (6.56) | -5.0 (10.71)
  SBP, conversion 2, 3 hours: number analyzed (Participants) | 5 | 9 | 12 | 7 | 6 | 4
  SBP, conversion 2, 3 hours | -12.0 (13.51) | -4.6 (11.64) | -3.3 (12.01) | 0.7 (14.13) | -5.0 (9.49) | -4.3 (8.81)
  SBP, conversion 2, 4 hours: number analyzed (Participants) | 4 | 4 | 10 | 5 | 6 | 4
  SBP, conversion 2, 4 hours | 1.0 (10.61) | -6.8 (4.27) | -2.6 (14.04) | 6.4 (4.04) | 0.3 (13.41) | -7.3 (5.56)
  SBP, conversion 2, 5 hours: number analyzed (Participants) | 2 | 3 | 6 | 3 | 3 | 1
  SBP, conversion 2, 5 hours | -9.0 (7.07) | -11.0 (11.36) | -0.5 (13.10) | 3.7 (9.45) | -18.0 (8.54) | 9.0 (NA) — only one participant was analyzed, hence SD was not calculated
  SBP, conversion 2, 6 hours: number analyzed (Participants) | 1 | 1 | 5 | 1 | 2 | 0
  SBP, conversion 2, 6 hours | -8.0 (NA) — only one participant was analyzed, hence SD was not calculated. | 3.0 (NA) — only one participant was analyzed, hence SD was not calculated. | -0.6 (14.84) | -7.0 (NA) — only one participant was analyzed, hence SD was not calculated. | -20.5 (7.78) |
  DBP, conversion 1, <30 minutes: number analyzed (Participants) | 1 | 0 | 1 | 1 | 0 | 0
  DBP, conversion 1, <30 minutes | -6.0 (NA) — only one participant was analyzed, hence SD was not calculated. |  | -2.0 (NA) — only one participant was analyzed, hence SD was not calculated. | -2.0 (NA) — only one participant was analyzed, hence SD was not calculated. |  |
  DBP, conversion 1, 1 hour: number analyzed (Participants) | 12 | 14 | 14 | 12 | 8 | 2
  DBP, conversion 1, 1 hour | -4.9 (6.69) | -4.7 (10.37) | -1.6 (9.46) | -1.5 (9.64) | -5.4 (8.55) | -5.0 (1.41)
  DBP, conversion 1, 2 hours: number analyzed (Participants) | 11 | 15 | 13 | 11 | 8 | 2
  DBP, conversion 1, 2 hours | -9.0 (13.59) | -2.9 (10.53) | -0.4 (7.32) | -4.8 (6.71) | -3.4 (7.25) | 6.0 (4.24)
  DBP, conversion 1, 3 hours: number analyzed (Participants) | 12 | 12 | 11 | 10 | 5 | 2
  DBP, conversion 1, 3 hours | -4.9 (10.89) | -1.9 (9.72) | -8.1 (11.26) | -9.2 (9.14) | -5.4 (7.96) | -5.0 (8.49)
  DBP, conversion 1, 4 hours: number analyzed (Participants) | 7 | 11 | 10 | 8 | 4 | 2
  DBP, conversion 1, 4 hours | -5.3 (6.82) | -9.7 (10.74) | -8.4 (8.41) | -5.1 (8.11) | -4.0 (10.89) | 4.0 (4.24)
  DBP, conversion 1, 5 hours: number analyzed (Participants) | 5 | 7 | 4 | 4 | 2 | 1
  DBP, conversion 1, 5 hours | -1.2 (2.28) | -8.4 (14.13) | -10.0 (9.42) | -5.8 (9.29) | -14.5 (9.19) | 0.0 (0.0)
  DBP, conversion 1, 6 hours: number analyzed (Participants) | 3 | 1 | 3 | 2 | 0 | 1
  DBP, conversion 1, 6 hours | -9.0 (4.36) | -23.0 (NA) — only one participant was analyzed, hence SD was not calculated. | -3.3 (2.08) | -6.0 (9.90) |  | 8.0 (NA) — only one participant was analyzed, hence SD was not calculated.
  DBP, conversion 2, <30 minutes: number analyzed (Participants) | 0 | 1 | 0 | 0 | 2 | 1
  DBP, conversion 2, <30 minutes |  | -10.0 (NA) — only one participant was analyzed, hence SD was not calculated. |  |  | -4.5 (0.71) | 20.0 (NA) — only one participant was analyzed, hence SD was not calculated.
  DBP, conversion 2, 1 hour: number analyzed (Participants) | 5 | 12 | 11 | 7 | 9 | 5
  DBP, conversion 2, 1 hour | -0.4 (12.70) | -5.1 (10.37) | -1.9 (8.50) | 0.9 (12.86) | 0.2 (8.97) | 3.8 (7.69)
  DBP, conversion 2, 2 hours: number analyzed (Participants) | 5 | 11 | 12 | 7 | 8 | 4
  DBP, conversion 2, 2 hours | 4.6 (12.42) | -9.6 (11.90) | -3.3 (11.19) | 0.9 (15.45) | -4.4 (8.62) | -10.5 (9.15)
  DBP, conversion 2, 3 hours: number analyzed (Participants) | 5 | 9 | 12 | 7 | 6 | 4
  DBP, conversion 2, 3 hours | 2.4 (20.42) | -5.8 (7.12) | -10.5 (14.16) | -1.4 (10.67) | -7.2 (5.71) | -4.5 (7.59)
  DBP, conversion 2, 4 hours: number analyzed (Participants) | 4 | 4 | 10 | 5 | 6 | 4
  DBP, conversion 2, 4 hours | 0.8 (17.11) | -8.3 (10.14) | -4.6 (17.66) | -1.0 (10.51) | -3.8 (7.19) | -7.8 (7.97)
  DBP, conversion 2, 5 hours: number analyzed (Participants) | 2 | 3 | 6 | 3 | 3 | 1
  DBP, conversion 2, 5 hours | -8.0 (0.00) | -2.3 (13.61) | -7.5 (13.71) | 2.0 (16.09) | -17.0 (5.20) | 8.0 (NA) — only one participant was analyzed, hence no data.
  DBP, conversion 2, 6 hours: number analyzed (Participants) | 1 | 1 | 5 | 1 | 2 | 0
  DBP, conversion 2, 6 hours | -7.0 (NA) — only one participant was analyzed, hence SD was not calculated. | -10.0 (NA) — only one participant was analyzed, hence SD was not calculated. | -5.8 (20.03) | -15.0 (NA) — only one participant was analyzed, hence SD was not calculated. | -15.0 (1.41) |

ADVERSE EVENTS:
Time Frame: Up to 5 weeks
Description: Conversion population was used. AEs and SAEs are also reported for participants who were included in pre and post conversion population. AEs were counted under the formulation the participant was taking, when the AE began. Hence, AEs data were reported formulation wise (Formulation A, B and C).
Arm/Group | Ropinirole Cohort A | Ropinirole Cohort B | Ropinirole Cohort C
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/53 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/52 | 0/53 | 0/30
Other Adverse Events (participants affected / at risk) | 37/52 | 38/53 | 19/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ropinirole Cohort A (N=52) | Ropinirole Cohort B (N=53) | Ropinirole Cohort C (N=30)
Palpitations (Cardiac disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ropinirole Cohort A (N=52) | Ropinirole Cohort B (N=53) | Ropinirole Cohort C (N=30)
Headache (Nervous system disorders) | 16 | 18 | 5
Nausea (Gastrointestinal disorders) | 10 | 15 | 9
Dizziness (Nervous system disorders) | 7 | 2 | 2
Somnolence (Nervous system disorders) | 4 | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 4 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Insomnia (Nervous system disorders) | 4 | 2 | 1
Nasopharyngitis (Infections and infestations) | 3 | 0 | 0
Restless legs syndrome (Musculoskeletal and connective tissue disorders) | 3 | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Fatigue (General disorders) | 2 | 3 | 1
Stomach discomfort (Gastrointestinal disorders) | 2 | 0 | 1
Paresthesia (Nervous system disorders) | 2 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 3 | 2
Hypertension (Vascular disorders) | 2 | 1 | 0
Influenza (Infections and infestations) | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 | 4 | 2
Vomiting (Gastrointestinal disorders) | 1 | 5 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 1
Hypoaesthesia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.